CLINICAL TRIAL: NCT05435066
Title: Cancer ORigin Epigenetics-Harbinger Health - Collection of Blood and Tissue Samples From Cancer and Non-Cancer Subjects for Validation of a Novel Blood-Based Multi-Cancer Screening Test
Brief Title: Development and Validation of Harbinger Health Test for Early Cancer Detection
Acronym: CORE-HH
Status: Completed | Type: Observational
Sponsor: Harbinger Health (Industry)
Responsible Party: Sponsor
Other Study IDs: HH-PRT-0001; Tissue 32 (Other: SCDI)
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: cancer; early detection; blood-based cancer screening; cfDNA; cancer diagnosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Tissue
  * Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm 1 - cancer group: Arm 1 - newly diagnosed cancer subjects
  Interventions: Diagnostic Test: Harbinger Health Test
- Arm 2 - non cancer group: Arm 2 - non-cancer subjects
  Interventions: Diagnostic Test: Harbinger Health Test

INTERVENTIONS:
Diagnostic Test: Harbinger Health Test — This trial will be used to test the ability of the Harbinger Health test to detect cancer using blood-based biomarkers in a large cohort of patients with cancer and matched non-cancer controls. The non-cancer controls will be followed for up to 1 year

SUMMARY:
This is a prospective, multi-center, observational study with a collection of biospecimens and clinical data from approximately 10,000 participants from up to 125 clinical network sites and locations in the United States. The objective of this study is to collect blood samples, tissue samples, and associated clinical data from participants with a variety of solid tumor and hematologic cancers and non-cancer participants for testing and the development of a screening test for early cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria - Both arms

Subjects must meet the following criteria in order to be included in the research study:

* Written or electronic informed consent
* Subject is 20 - 79 years of age at the time of signature of the informed consent form (ICF)
* Male or female subjects

Inclusion Criteria Arm 1 - Cancer Subjects Arm 1 subjects enrolled in the study must meet the following inclusion criteria.

* A confirmed diagnosis or high suspicion of cancer (stage I to IV solid cancer or hematologic cancer) by imaging within 180 days prior to enrollment; not to include myelodysplastic and myeloproliferative syndromes
* Subject's cancer diagnosis is based upon assessment of a pathological specimen or high suspicion of cancer by imaging
* Subject's cancer is treatment-naïve

Inclusion Criteria Arm 2 - Non-Cancer Subjects (All Cohorts)

Arm 2 subjects enrolled in the study must meet the following inclusion criteria:

* Subject's health permits participation and the subject is not suspected of having cancer based on provider assessment.
* The subject was not diagnosed with cancer or received cancer treatment within the last 5 years (persons with completely resected ductal carcinoma in-situ or non-melanoma skin cancer are permitted).

Part 1B Only :

- Subject has no known current cancer and has 1 of the follow conditions:

o An Advanced Adenoma (AA) of the gastrointestinal tract as defined as an adenoma that is ≤10mm in size Subjects with any one of the criteria would be eligible High grade displasia or ≥10 adenoma: any size Tubulovillous adenoma, any size Tubular adenoma ≥10mm Traditional serrated adenoma ≥10mm

Exclusion Criteria:

Subject self-reporting OR available medical records at the time of screening are acceptable for assessment of all exclusion criteria.

Exclusion Criteria - Both arms

Subjects who meet any of the following criteria will be excluded from study entry:

* Subject is suffering from any febrile illness defined as a temperature >101.5°F within the last 48 hrs.
* Subject is pregnant (by self-report of pregnancy status).

Exclusion Criteria Arm 1 - Cancer Subjects

Subjects who meet any of the following criteria will be excluded from study entry:

* Subject with a prior history of cancer within 5 years will not be allowed to participate in the study
* More than 1 active cancer diagnosis (ie. a subject presenting with recurrent breast cancer and newly diagnosed lung cancer would be excluded; subject with prior (>5 years ago) treated breast cancer without recurrence and presenting with newly diagnosed lung cancer would be eligible).
* Subject is currently receiving, or has in the past received, any of the following definitive therapies to treat their current cancer:

  * Surgical treatment, surgical removal, or surgical management of the cancer beyond that required to establish the cancer diagnosis. Surgical or biopsy procedures that remove more tissue than required to establish the cancer diagnosis, or that were performed to manage symptoms or initiate cancer treatment prior to blood sample collection will be considered 'definitive' and are not permissible regardless of the residual tumor mass remaining in the subject.
  * Chemotherapy (local, regional, or systemic) including chemoembolization targeted therapy;
  * Immunotherapy including cancer vaccines;
  * Hormone therapy; or
  * Radiation therapy (a single dose of palliative radiation prior to study start is allowed).
* The subject is a recipient of an organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Subject who has undergone a bowel preparation for a gastrointestinal malignancy within 3 days of an anticipated blood draw.

Exclusion Criteria Arm 2 - Non-cancer Subjects

Subjects who meet any of the following criteria will be excluded from study entry:

- The subject is the recipient of an organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed cancer subjects and non-cancer subjects
Sampling Method: Non-Probability Sample
Enrollment: 8038 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Detection of cancer or non-cancer using Harbinger Test | Up to 12 months
  Analyze Subject's cfDNA from blood samples for "cancer" or "non-cancer" signals using the Harbinger Health test, and compare results of the test to clinical diagnosis
Performance for specific cancer types using Harbinger Test | Up to 12 months
  Sub-analysis by clinical diagnosis of cancer type (e.g. Breast cancer) to determine how well the Harbinger Health test detects specific tumor types
Identify the correct tumor type by Harbinger Test | Up to 12 months
  Analyze Subject's cfDNA from blood samples to accurately identify specific tumor types (e.g. Breast cancer) using the Harbinger Health test, by comparing results of the test to clinical diagnosis

SECONDARY OUTCOMES:
Evaluate performance of the Harbinger Health Test by tumor stage | Up to 12 months
  Assess Harbinger Health test performance with repeat of primary subgroup analysis through Tumor Stage within Cancer Type.
Evaluate performance of the Harbinger Health Test to discriminate hyperplasia Advanced Adenoma. | Up to 12 months
  Assess Harbinger Health test performance by repeat of Primary with Subgroup Analysis of Non-Cancer vs. Hyperplasia (Advanced Adenoma).

CONTACTS AND LOCATIONS:
Overall Officials: Dax Kurbegov, MD, Study Chair — Sarah Cannon; Hutan Ashrafian, MD MBA PhD, Study Director — Harbinger Health; Luke Pike, MD DPhil, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (125):
- United States (125):
  - Southern Cancer Center, Daphne, Alabama
  - Alaska Oncology and Hematology, LLC, Anchorage, Alaska
  - Alaska Womens Cancer Care, Anchorage, Alaska
  - Arizona Oncology Associates HAL, Prescott Valley, Arizona
  - Pacific Cancer Medical Center, Anaheim, California
  - Central California ENT Medical Group, Fresno, California
  - South Coast Gynecologic Oncology, Inc, San Diego, California
  - South Coast Gynecologic Oncology, INC, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Gynecologic Oncology Associates, Torrance, California
  - Colorado Primary Health Care, Littleton, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Central Florida Pulmonary Group - Altamonte Springs, Altamonte Springs, Florida
  - ENT and Allergy Associates of Florida, LLC, Boca Raton, Florida
  - Plastic Surgery Specialists of Boca Raton, Boca Raton, Florida
  - South Florida Center for Gynecologic Oncology, Boca Raton, Florida
  - Urology Center of South Florida, Boynton Beach, Florida
  - Advanced Cancer Surgery and Digestive Health, Boynton Beach, Florida
  - ENT and Allergy Associates of Florida, LLC, Brandon, Florida
  - Zoyla Almedia, MD PA, Coconut Creek, Florida
  - ENT and Allergy Associates of Florida, LLC, Ft. Pierce, Florida
  - Stuart Oncology Associates, Ft. Pierce, Florida
  - I.H.S. Health, Kissimmee, Florida
  - ENT and Allergy Associates of Florida, LLC - Okeechobee, Okeechobee, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Central Florida Pulmonary Group - Dylan Loren Cir, Orlando, Florida
  - Cancer Care Centers of Brevard, Palm Bay, Florida
  - ENT and Allergy Associates of Florida, LLC, Palm Beach Gardens, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - ENT and Allergy Associates of Florida, LLC, Plantation, Florida
  - ENT and Allergy Associates of Florida, LLC, Port Saint Lucie, Florida
  - Stuart Oncology Associates, Port Saint Lucie, Florida
  - Stuart Oncology Associates, Stuart, Florida
  - ENT and Allergy Associates of Florida, LLC, Wesley Chapel, Florida
  - ENT and Allergy Associates of Florida, LLC, West Palm Beach, Florida
  - Advanced Urology - John's Creek, Johns Creek, Georgia
  - Advanced Urology - Lawrenceville, Lawrenceville, Georgia
  - Advanced Urology - Marietta, Marietta, Georgia
  - Advanced Urology - Rosewell, Roswell, Georgia
  - Advanced Urology - Snellville, Snellville, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Hem/Onc of the North Shore, Skokie, Illinois
  - Evansville Surgical Associates-Mary Street, Evansville, Indiana
  - Evansville Surgical Associates-Mary's Drive, Evansville, Indiana
  - Evansville Surgical Associates-Gateway Boulevard, Newburgh, Indiana
  - Mission Cancer and Blood, Des Moines, Iowa
  - Wichita Urology Group - W. 21st Street, Wichita, Kansas
  - Wichita Urology Group- P.A. - 2077 N. Webb Road, Wichita, Kansas
  - Breast Care Specialists, Wichita, Kansas
  - Kansas Surgery & Recovery Center, Wichita, Kansas
  - Wichita Urology Group- 2626 Webb Road, Wichita, Kansas
  - Northlake Gastroenterology Associates, Hammond, Louisiana
  - Maryland Oncology Hematology, Columbia, Maryland
  - Comprehensive Urology - Farmington Hills, Farmington Hills, Michigan
  - Comprehensive Urology - Novi, Novi, Michigan
  - Comprehensive Urology - Roseville, Roseville, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Comprehensive Urology - Royal Oak, Royal Oak, Michigan
  - Comprehensive Urology - Sterling Heights, Sterling Heights, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Somnos Clinical Research, Lincoln, Nebraska
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - New Jersey Cancer Care, Belleville, New Jersey
  - New Jersey Hematology Oncology Associates, Brick, New Jersey
  - Surgical Specialists of New York - Jersey City, Jersey City, New Jersey
  - Oncology Hematology Specialists, Mountain Lakes, New Jersey
  - Center of Dermatology and Skin Surgery, LLC, Paramus, New Jersey
  - Women's Cancer Care Associates LLC, Albany, New York
  - Surgical Specialists of NY - Astoria, Astoria, New York
  - New York Gastroenterology Associates - Pierrepont, Brooklyn, New York
  - Gardith Joseph Medical P.C. Quality Cancer Care, Brooklyn, New York
  - Vantage Medical Associates, Brooklyn, New York
  - Associated Gastroenterologists of Central New York - Camillus, Camillus, New York
  - Associated Gastroenterologists of Central New York - Syracuse, East Syracuse, New York
  - Vantage Medical Associates, Far Rockaway, New York
  - Associated Gastroenterologists of Central New York - Fayetteville, Fayetteville, New York
  - Hudson Valley Cancer Center - Fishkill, Fishkill, New York
  - Advanced Urology Centers of NY, Lake Success, New York
  - Gastroenterology Oncology Associates, Liverpool, New York
  - New York Gastroenterology Associates - Columbus Ave, New York, New York
  - New York Gastroenterology Associates - 86th Street, New York, New York
  - New York Gastroenterology Associates - E 79th St, New York, New York
  - New York Gastroenterology Associates - 5th Ave, New York, New York
  - Surgical Specialists of NY - New York City, New York, New York
  - Advanced Radiation Oncology Services, Nyack, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Hudson Valley Cancer Center - Poughkeepsie, Poughkeepsie, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Hirschfeld Oncology, The Bronx, New York
  - Westmed Medical Group, Woodmere, New York
  - Hudson Valley Cancer Center - Yorktown Heights, Yorktown Heights, New York
  - Dayton Physicians Network, Dayton, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - Northwest Cancer Specialists-, Portland, Oregon
  - Eastern Pennsylvania Gastroenterology & Liver Specialists, LLC, Allentown, Pennsylvania
  - Blair Gastroenterology Associates, Altoona, Pennsylvania
  - Consultants in Medical Oncology & Hematology, Broomall, Pennsylvania
  - Pulmonology Associates INC., Wynnewood, Pennsylvania
  - Pulmonology Associates INC, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - GIA Clinical Trials, LLC, Knoxville, Tennessee
  - Advantage Clinical Research, Nashville, Tennessee
  - HCA research Institute, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Texas Oncology - West Texas, Amarillo, Texas
  - Texas Oncology - Gulf Coast, Beaumont, Texas
  - Texas Oncology - Dallas, Dallas, Texas
  - Texas Oncology - Presbyterian Cancer Center Dallas, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Fort Worth, Fort Worth, Texas
  - Houston Digestive Diseases Consultants, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - Northeast Texas Cancer and Research, McKinney, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - Plano West, Plano, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Center for Digestive Disease, Shenandoah, Texas
  - Texas Oncology - Northeast Texas Cancer and Research, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Shenandoah Oncology, Winchester, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington